CLINICAL TRIAL: NCT05149586
Title: Principle Investigator
Brief Title: Impact of Low Dose Ketamine Infusion in Septic Patient on Non-invasive Estimators of ICP
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Essamedin Mamdouh Negm, principal investigator, Zagazig University
Other Study IDs: 6928-6-9-2021
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Intracranial Pressure Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe sepsis is a major healthcare problem with a reported incidence of 1-2% in all hospitalizations. It is a major cause of death in the intensive care units worldwide and is the second leading cause of death in noncoronary intensive care unit patients. Mortality remains high at 30-50% despite a better understanding of sepsis pathophysiology and improved advanced care in the past decade .

Sedation and analgesia in the intensive care unit (ICU) for patients with sepsis and tenuous hemodynamics can be challenging. Opioids and benzodiazepines can contribute to the pathophysiology of shock by exacerbating poor tissue perfusion through reduced cardiac contractility, and increased vasodilation as well as reducing the respiratory drive .

Sedation and analgesia management are both integral components of care in the intensive care unit (ICU). Although benzodiazepines have been the mainstay therapy for sedation in critically ill patients, their use has declined in recent years, with favoring of nonbenzodiazepines,such as propofol and dexmedetomidine .

A noticeable interest in ketamine infusion for sedation management in critically ill patients has developed among critical care physicians . The 2018 Pain, Agitation/ sedation, Delirium, Immobility, and Sleep disruption (PADIS) guideline suggested low-dose ketamine as an adjunct to opioid therapy for reducing opioid consumption in post-surgical adults admitted to the ICU .

Ketamine affects many pathways leading to inflammation cascade during sepsis. First, ketamine has an immunosuppressive effect on immune cells such as NK cell cytotoxic activity, neutrophil adhesion to endothelium, and chemotactic activity of neutrophils. Second, ketamine decreases Toll-like receptor expression, nuclear factorkB activity, and Raf/Raf cascade. Third, ketamine suppresses cytokines, superoxide, and nitric oxide productions, and reduces the mitochondrial membrane potential in macrophages. Finally, ketamine prevents the alteration of immune function in patients early after a major surgery, and increases survival in rats with sepsis .

Cerebral perfusion pressure (CPP) was compromised only in the patients with pre-existing intracranial hypertension and obstruction to the flow of cerebral spinal fluid. This has, however, led to the persistent belief that ketamine is contraindicated in patients with traumatic head injuries. Studies done subsequently have shown, however, that the effects of ketamine on cerebral haemodynamics and ICP are in fact variable and depend on both the presence of additional anaesthetic agents and PaCO2 values . Meta-analysis also suggests that Ketamine does not increase ICP and provides favorable hemodynamics . Meta analysis has shown that when ketamine is used in the presence of controlled ventilation, in conjunction with anaesthetics which reduce cerebral metabolism such as GABA receptor agonists, ICP is not increased.

The gold standard technique for ICP measurement is an intraventricular catheter[10]; however, this method is invasive and can have complications . Non-invasive ICP (nICP) measurement is a promising technique, still under development in adult and pediatric population .Optic nerve sheath diameter (ONSD) measurement using ocular ultrasonography is a safe, quick, reliable and reproducible technique for the assessment of ICP . Transcranial Doppler Ultrasonography (TCD) can also non-invasively assess ICP and CPP. Increased ICP produces characteristic changes in cerebral blood flow velocity (FV) waveform that can be assessed by decreases in the diastolic FV and increases in the pulsatility index (PI=systolic FV - diastolic FV) / mean FV) and several methods TCD derived have been proposed to assess non invasively ICP, showing good performance .

Sepsis-associated encephalopathy (SAE) usually manifests as sleep awakening cycle disturbance, cognitive impairment, delirium, and coma . Considering that brain edema secondary to SAE is one of the complications and causes of death in patients with sepsis, early detection of intracranial hypertension (ICH) is of great significance for timely intervention and improved prognosis. However, most patients with sepsis without intracranial infection have no indications for invasive intracranial pressure (ICP) monitoring; thus, non-invasive ICP monitoring was selected .

Therefore, in patients without invasive ICP monitoring, nICP methods may be useful for determining if ketamine infusion in septic patient will cause a pathological increase in ICP.

ELIGIBILITY:
Inclusion Criteria:

1. Patient acceptance (if conscious)
2. Age >18years.
3. Sex: both.
4. septic patient.

Exclusion Criteria:

1. Patient refusal
2. Inflammatory lesions of the optic nerve itself (optic neuritis)
3. Trauma to eye like rupture globe
4. Glaucoma and optic atrophy
5. History of previous intracranial surgery or spinal cord disease.
6. Pregnant patients
7. known allergy to ketamine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: septic patient admitted to intensive care units at zagazig university hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
1- To compare the ICP monitoring after ketamine infusion in septic patient | 4 months
  To evaluate ICP monitoring parameters before and after ketamine infusion in septic patient (changes in ICP parameters)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided